CLINICAL TRIAL: NCT04579926
Title: PINPOINT: Gaming Technology to Engage Adolescent Sickle Cell Patients in Precision Pain Phase II
Brief Title: PINPOINT: Gaming Technology for SCD Pain
Acronym: Pinpoint II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); HPC International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 322; R44MD010746-02 (NIH)
Record Dates: First submitted 2020-09-17; First posted 2020-10-08 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia in Children; Sickle Cell Thalassemia; Sickle Cell SC Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Randomized step wedge design with multiple baselines. Parents and adolescents were enrolled as dyads. Only adolescents received the intervention and will be reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pinpoint App (Experimental): Tablet and smartphone application.
  Interventions: Other: Pinpoint app

INTERVENTIONS:
Other: Pinpoint app — Tablet and smartphone app with pain assessment and communication education, and pain assessment tool.

SUMMARY:
Sickle cell disease (SCD) is a common genetic disorder characterized by episodes of pain, yet programs to assist SCD adolescents with better identification and communication about pain are lacking. Research shows that interactive gaming technology can enhance adolescents' learning, and can be especially effective in delivering health-related messages and tools to improve self-care. Pinpoint is an interactive gaming app that will be tested in a Phase II project to determine whether the app assists SCD teens with improving their communication and identification skills for pain self-report.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is the most common inherited blood disorder in the U.S. and disproportionately affects African Americans and Hispanics. Approximately, 1,000 U.S. children are born with SCD annually. SCD results from abnormal hemoglobin and causes red blood cells (RBCs) to become misshaped ("sickle-shaped"). Sickled cells can block the flow of blood in small arteries causing tissue and organ damage and other life-threatening comorbidities. SCD complications can be serious and have a significant impact upon well-being and quality of life. Pain is the hallmark symptom associated with SCD, and is the most common clinical problem seen in children and the number one cause of SCD-related hospital admissions. If left untreated, these painful episodes can result in morbidity and mortality. Accurate assessment of pain specifiers (type, frequency, and intensity of pain) can help with ameliorating pain quickly and effectively. Despite children being accurate self-reporters of their pain, strategies which are effective and engaging to assist with pain identification and communication of pain are lacking. In a Phase I SBIR, the investigator's team examined the feasibility and acceptability of a gamified tablet application (Pinpoint) intended to encourage teens to talk about and assess their SCD pain. The Phase I specific aims were : (1) work with an Expert Advisory Board (EAB) of experts to develop a new pain assessment tool (PAT) to engage adolescent SCD patients, improve pain specification by patients, and improve pain management by clinicians; (2) conduct cognitive interviews and focus groups with 13-17 year old SCD patients to guide and refine development of app content, design, and aesthetics to fully develop a functioning prototype; (3) conduct usability testing with 13-17 year old SCD patients to assess functionality, navigation, and satisfaction; (4) conduct cognitive interviews with medical providers to provide input on app content, perceived barriers to use, and its potential for clinical use and integration to inform future implementation; and (5) develop a specifications document to outline the Phase II development plan. Deliverables were met and feasibility was confirmed by the EAB. The proposed Phase II project will (1) develop a fully programmed, interactive Pinpoint app consisting of modules to address pain identification and communication; (2) conduct usability testing of Pinpoint to evaluate the user interface, ease of use, and perceived barriers in order to optimize the app prior to large scale evaluation (n=14); and (3) test the full app with 13-17 year olds with SCD (n=100) using a randomized step wedge design to evaluate changes in (a) knowledge acquisition for communicating about pain and types of pain; (b) the Pain Assessment; (c) SCD general knowledge and self-efficacy; (d) family cohesion; and (e) app usage. Overall, the proposed project has the potential to significantly impact the health of SCD teens by providing important skill acquisition for communicating about and identifying pain. This project is innovative and timely. Pinpoint will be the first app to identify and translate specific pain types for SCD into a gamified app using applied gamification principles.

ELIGIBILITY:
Inclusion Criteria:

* Be 13-17 years of age
* Be diagnosed with sickle cell disease
* Able to read and speak English
* Able to assent to participate

Exclusion Criteria:

* Not 13-17 years of age
* Not diagnosed with sickle cell disease
* Unable to read and speak English
* Unable to assent to participate

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Myers, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Klein Buendel, Inc., Golden, Colorado
  - Hilton Publishing Company, Munster, Indiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Pinpoint App: Tablet and smartphone application.
  Pinpoint app: Tablet and smartphone app with pain assessment and communication education, and pain assessment tool.
  Parent-adolescent dyads were randomized, but only adolescents received the intervention and were assessed for outcome measures.
Period: Overall Study
Arm/Group | Pinpoint App
Started | 24
Parents | 24
Adolescents | 24
Completed (For the stepped wedge design, n=18 were instructed to complete 0 week, 4 week, 8 week, and 12 week. n=6 were instructed to complete 0 week, 4 week, 8 week, and 12 week, and 16 week surveys.) | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adolescents and parents were randomized as dyads, but the intervention was designed for adolescents and only adolescents were included in analyses. All outcome measures are based on adolescents.
Arm/Group | Pinpoint App
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.75 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Sickle Cell Self-efficacy Scale Reported by Adolescents
Description: Sickle Cell Disease (SCD) self-efficacy: This instrument, used to assess self-efficacy in adolescents with SCD, is comprised of 9 questions measuring participants' perceptions of their ability to function on a day-to-day basis and to manage SCD symptoms (e.g., pain). The instrument is reliable and valid for assessing adolescents' self-efficacy for engaging successfully in day-to-day activities despite having SCD. Responses from individual items are summed to give an overall score. Higher scores indicate greater self-efficacy. Range = 0-45 (min=10 max=45).
Time Frame: baseline
Population: adolescents
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pinpoint App
Number analyzed (Participants) | 24
units on a scale | 34.6 (8.3)

2. Primary Outcome: Sickle Cell Self-efficacy Scale Reported by Adolescents
Description: Sickle Cell Disease (SCD) self-efficacy: This instrument, used to assess self-efficacy in adolescents with SCD, is comprised of 9 questions measuring participants' perceptions of their ability to function on a day-to-day basis and to manage SCD symptoms (e.g., pain). The instrument is reliable and valid for assessing adolescents' self-efficacy for engaging successfully in day-to-day activities despite having SCD. Responses from individual items are summed to give an overall score, with higher scores indicating greater self-efficacy. Range = 0-45 (min= 9; max = 45).
Time Frame: 4-weeks
Population: adolescents
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pinpoint App
Number analyzed (Participants) | 24
units on a scale | 35.8 (8.3)

3. Primary Outcome: Sickle Cell Self-efficacy Scale Reported by Adolescents
Description: Sickle Cell Disease (SCD) self-efficacy: This instrument, used to assess self-efficacy in adolescents with SCD, is comprised of 9 questions measuring participants' perceptions of their ability to function on a day-to-day basis and to manage SCD symptoms (e.g., pain). The instrument is reliable and valid for assessing adolescents' self-efficacy for engaging successfully in day-to-day activities despite having SCD. Responses from individual items are summed to give an overall score. Higher scores indicate greater self-efficacy. Range = 0-45 (min= 24 max=45).
Time Frame: 8-weeks
Population: adolescents
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pinpoint App
Number analyzed (Participants) | 24
units on a scale | 37.4 (5.9)

4. Primary Outcome: Sickle Cell Self-efficacy Scale Reported by Adolescents
Description: Sickle Cell Disease (SCD) self-efficacy: This instrument, used to assess self-efficacy in adolescents with SCD, is comprised of 9 questions measuring participants' perceptions of their ability to function on a day-to-day basis and to manage SCD symptoms (e.g., pain). The instrument is reliable and valid for assessing adolescents' self-efficacy for engaging successfully in day-to-day activities despite having SCD. Responses from individual items are summed to give an overall score, with higher scores indicating greater self-efficacy. Range = 0-45 (min=26 max=45).
Time Frame: 12-weeks
Population: adolescents
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pinpoint App
Number analyzed (Participants) | 24
units on a scale | 38.9 (6.5)

5. Primary Outcome: Sickle Cell Self-efficacy Scale
Description: Sickle Cell Disease (SCD) self-efficacy: This instrument, used to assess self-efficacy in adolescents with SCD, is comprised of 9 questions measuring participants' perceptions of their ability to function on a day-to-day basis and to manage SCD symptoms (e.g., pain). The instrument is reliable and valid for assessing adolescents' self-efficacy for engaging successfully in day-to-day activities despite having SCD. Responses from individual items are summed to give an overall score, with higher scores indicating greater self-efficacy. Range = 0-45 (min=18 max=45).
Time Frame: 16-weeks
Population: adolescents eligible from stepped wedge design
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pinpoint App
Number analyzed (Participants) | 6
units on a scale | 39.0 (10.5)

6. Secondary Outcome: System Usability Scale (SUS)
Description: Technology acceptability: The System Usability Scale (SUS) is a reliable tool for measuring the usability of technologies. It consists of a 10-item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking. Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average. Range = 37.5-100
Time Frame: final posttest (either 12-weeks or 16-weeks, per stepped wedge design)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pinpoint App
Number analyzed (Participants) | 23
units on a scale | 72.5 (19.1)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Pinpoint App
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT04579926/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT04579926/ICF_001.pdf